CLINICAL TRIAL: NCT04154215
Title: FDG Metabolism in Dementia With Lewy Body (DLB) Patients as Indicated by PET Dynamic Acquisition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0516-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia with Lewy Body (DLB) patients (Experimental)
  Interventions: Diagnostic Test: PET-CT FDG brain scan

INTERVENTIONS:
Diagnostic Test: PET-CT FDG brain scan — Scans will be performed in Discovery MI PET/CT scanner (by GE). Dynamic FDG PET scan start immediately after a bolus injection of 18F-FDG (0.1 mCi/kg) 5. Dynamic PET scan protocol of 30 min will be follow by a static scan protocol with a duration of 8 min combined with a low dose CT scan.
  The radiation exposure of the patients is equal to the radiation exposure during the routine PET-CT FDG brain scan. The only discomfort to the patient is a longer scan duration.
  After the scan is concluded the patient will be released with no restrictions. Each of the acquired PET images will undergo visual assessment. In addition, quantification of the image data using Standardized Uptake Values (SUV) and kinetic model. The correlation between the clinical information, visual assessment and quantitative parameters will be tested. Sensitivity and accuracy of the quantification methods will be calculated.

SUMMARY:
Dementia with Lewy Body (DLB) is a common neurodegenerative disorder responsible to 15%-20% of the dementia cases in the elderly population.

Dementia with Lewy Body (DLB) is a common neurodegenerative disorder responsible to 15%-20% of the dementia cases in the elderly population . This disorder belongs to the family of synucleinopathies, which are diseases characterized by the abnormal accumulation of the protein α-synuclein (α-syn) in neuronal and non-neuronal cells in the brain. The clinical symptoms of DLB include dementia with the presence of fluctuations in attention or alertness, recurrent visual hallucinations, spontaneous extrapyramidal motor features and REM sleep behavior disorder (RBD). Supportive clinical symptoms are severe sensitivity to antipsychotic agents, postural instability, repeated falls, syncope or other transient episodes of unresponsiveness, severe autonomic dysfunction e.g. constipation, orthostatic hypotension, urinary incontinence, hypersomnia, hyposmia, hallucinations in other modalities, systematized delusions, apathy, anxiety and depression. DLB differs from PD by the order of appearance of clinical symptoms.

The diagnosis of DLB requires in addition to the clinical symptoms the existence biomarkers indicating the pathology. It is important to note that due to the complexity of DLB diagnosis, mainly due to the similarity of this syndrome to other dementia conditions, more than one biomarker is required to identify DLB [6]. The biomarkers contain indicative biomarkers and supportive biomarkers. Indicative biomarkers include a. Assessment of the integrity of dopaminergic system by either F-DOPA Positron Emission Tomography (PET) or by Ioflupane 123I (DaT) Single Photon Emission Tomography (SPECT) scans. b. Abnormal (low uptake) MIBG myocardial scintigraphy. c. Polysomnographic confirmation of REM sleep without atonia.

Supportive biomarkers are: a. MRI/CT scans showing neuronal structural modifications with relative preservation of medial temporal lobe structures. b. Generalized low uptake on SPECT/PET perfusion/metabolism scan with reduced occipital activity +/- the cingulate island sign on 18F-fludeoxyglucose (FDG) PET imaging. c. Prominent posterior slow wave activity on EEG with periodic fluctuations in the pre-alpha/theta range.

Biochemical biomarkers from the blood and spinal fluid were also investigated. These biomarkers include measurement of levels of Amyloid β, tau, and phospho-tau measurements. However, they do not allow differentiation between DLB and AD. α-syn was not proven as a biomarker.

DETAILED DESCRIPTION:
The purpose of this research is to assess whether dynamic FDG-PET scans and quantitative analysis of the these scans can give a more accurate and sensitive information regarding the DLB brain glucose metabolism which in turn may give better insight about DLB mechanism and allow better assessment of the disease.

Glucose metabolism in the brains of DLB patients is characterized by a pattern of bilateral parietal and posterior temporal hypometabolism with specific occipital hypo metabolic signature [9]. The use of FDG-PET scans allows the mapping of the topographic hypo metabolic view of the brain in different stages of the DLB condition. These metabolic maps, in turn, can be used both for diagnostic purposes as well as for research of the DLB mechanism [10] [11]. FDG is also a modality assisting in the differentiation between AD, PD and DLB [12]. To notice, the disadvantage of the FDG-PET scans is the lack of quantification. Visually analysis of brain FDG metabolism without quantitative analysis is limiting its use as a biomarker and the diagnostic accuracy and sensitivity of the scan. This is the main reason why it is considered only a supportive biomarker [9].

In these study the investigators will investigate the utilization of dynamic FDG PET scans in order to track in more close and precise way the path of the glucose metabolism in the brain. In addition, the investigators would like to use the dynamic scans to perform quantification of the FDG distribution in the brain in order to show the advantage of the quantification in the diagnostic process.

ELIGIBILITY:
Inclusion Criteria:

1. A cohort of healthy patients with no symptoms or family history of DLB will be tested as control group.
2. Healthy asymptomatic patients with first-degree relatives of DLB patients.
3. DLB patients that went through comprehensive neuropsychological assessments and were confirmed as suffering from DLB.

Exclusion Criteria:

1. Age <18.
2. Pregnant or breath feeding patients.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-14 (Estimated); Primary Completion 2020-01-14 (Estimated); Study Completion 2021-12-14 (Estimated)

PRIMARY OUTCOMES:
number of patients that have shown the tracer time activity curve between healthy, DLB and AD patients for differential diagnosis. | 1 year

IPD SHARING:
Plan to Share IPD: Undecided